CLINICAL TRIAL: NCT01706549
Title: Chronic Pain After Hysterectomy, Qualitative Analysis of Pain and Its Impact on Quality of Life
Brief Title: Clinical Analysis of Pain After Hysterectomy
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R11190
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Postoperative Pain
Keywords: Chronic pain; Hysterectomy; Quality of life
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Posthysterectomy pain: Observational study on posthysterectomy pain

SUMMARY:
Patients undergone either laparoscopic or vaginal hysterectomy will called for a clinical examination 1-3 years after surgery, if they suffer from pain 6 months after surgery. The aims of the study are:

1. to reveal whether the pain is postsurgical in nature, or if there are any other reasons for the pain.
2. to reveal the type of pain, neuropathic, nociceptive or idiopathic.
3. to reveal the impact of pain on quality of life.

DETAILED DESCRIPTION:
Patients undergone either laparoscopic or vaginal hysterectomy will called for a clinical examination 1-3 years after surgery, if they suffer from pain 6 months after surgery. All patients were treated in Pirkanmaa District Hospital and the anesthesia was either propofol-infusion or sevoflurane gas with remifentanil-infusion.

6months after the surgery, questionnaires about pelvic pain were sent to the patients. Patients still having pain at that time, were invited for detailed sensory and gynecological examinations.

ELIGIBILITY:
Inclusion Criteria:

* hysterectomy 1-3 years previously
* suffering from pain 6months postsurgically

Exclusion Criteria:

-

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergone hysterectomy for 1-3 years previously and suffering from persistent pain 6 months after surgery. The patients are invited to participate in this study, if they have participated in previous studies "Sevoflurane, Propofol, Postoperative pain" by Yli-Hankala and Pokkinen and study:" Vaginal hysterectomy, laparoscopic hysterectomy, postoperative pain" by Yli-Hankala and Pokkinen.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satu Pokkinen, MD, Principal Investigator — Tampere University Hospital; Maija-Liisa Kalliomäki, MD, PhD, Study Director — Tampere University Hospital; Kari Nieminen, MD, Doc, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2012-December 2013. Patients recruited from previous studies. Clinical evaluation at the Hospital on the basis of volunteering.
Groups:
- Posthysterectomy Pain: Observational study on posthysterectomy pain. Participants recruited from previous studies. Recruitment completed.
Period: Overall Study
Arm/Group | Posthysterectomy Pain
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients undergone hysterectomy and reportteri to have SUFFERED from pain 6 months postoperatively and volunteered for a clinical examination.
Groups:
- Postoperative Pain: Observational study on posthysterectomy pain
Arm/Group | Postoperative Pain
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51 (6.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 1
Gender [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Region of Enrollment [Number; unit: participants]
  Finland | 16
Quality of life (SF-36) [Mean (Standard Deviation); unit: units on a scale] — All dimensions are mean of points from 0-100, where 100 is the best score. Getting 0 points equals to poor performance.
  units on a scale
    Physical Functioning | 76.9 (29.2)
    Role Physical | 57.8 (45.7)
    Role Emotional | 54.1 (43.9)
    Vitality | 55.3 (24.8)
    Mental health | 70.0 (18.2)
    Social Functioning | 70.6 (26.8)
    Bodily Pain | 65.5 (29.2)
    General health | 56.8 (20.1)

OUTCOME MEASURES:

1. Primary Outcome: Type of Chronic Pain After Hysterectomy
Description: Number of participants with probable neuropathic, possible neuropathic, pain had subsided and other type of pain.
Time Frame: 1-3 years after hysterectomy
Population: Women undergone hysterectomy previously and reported having pain at the site of surgery six months after surgery
Measure: Number; unit: participants
Arm/Group | Posthysterectomy Pain
Number analyzed (Participants) | 16
participants
  Probable neuropathic pain | 5
  Possible neuropathic pain | 4
  Subsided pain | 6
  Other type of pain | 1

2. Secondary Outcome: Quality of Life After Hysterectomy
Description: Quality of life as measured by the SF-36, which consists of 8 scales.
Time Frame: 1-3 years after hysterectomy
Reporting Status: Not Posted

3. Secondary Outcome: Is the Pain Due to Hysterectomy?
Description: Number of patients having posthysterectomy pain versus other pain
Time Frame: 1-3 years
Measure: Number; unit: participants
Arm/Group | Posthysterectomy Pain
Number analyzed (Participants) | 16
participants | 15

ADVERSE EVENTS:
Time Frame: May 11th 2012-November 15th 2013
Description: This was an observational study, thus no adverse events were anticipated.
Groups:
- Posthysterectomy Pain: This was an observational study, thus no adverse events were collected.
Arm/Group | Posthysterectomy Pain
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Low participation rate. Inadequate filling of questionnaires. Time from surgery to clinical examination varied from 10 to 44 months. No preoperative quality of life measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes